CLINICAL TRIAL: NCT03302520
Title: Comparison of Fusion Rate and Clinical Results Between Bioactive Glass Ceramics Spacer With PEEK Cages in Posterior Lumbar Interbody Fusion: A Prospective, Randomized Controlled Non-inferiority Trial
Brief Title: Comparison of Bioactive Glass Ceramics Spacer and PEEK Cages in Posterior Lumbar Interbody Fusion: A Prospective, RCT
Acronym: Novomax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nvmax_001
Record Dates: First submitted 2017-09-21; First posted 2017-10-05 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Degenerative Lumbar Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novomax (Experimental): Novomax(R) ceramic glass spacer for interbody fusion
  Interventions: Device: NovoMax, BioAlpha Inc, Seong-nam, Korea
- PEEK cage (Active Comparator): PEEK cage for interbody fusion
  Interventions: Device: PEEK cage

INTERVENTIONS:
Device: NovoMax, BioAlpha Inc, Seong-nam, Korea — CaO-SiO2-P2O5-B2O3 glass ceramics spacer
  Arms: Novomax
Device: PEEK cage — PEEK cage
  Arms: PEEK cage

SUMMARY:
The authors aimed to compare the clinical efficacy and safety of CaO-SiO2-P2O5-B2O3 glass ceramics with PEEK cage that is widely used for posterior lumbar interbody fusion (PLIF) surgery in the clinical field.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 30 and 80
* patients who required one-level PLIF between L1 and S1 among those who required an extensive laminectomy or facetectomy to correct severe disc extrusion or severe spinal stenosis or those who required PLIF due to grade I or II spondylolisthesis
* those who (only if a signature was obtainable), or whose legal guardian, fully understood the clinical trial details and signed the informed consent form.

Exclusion Criteria:

* osteoporosis patients with average T-scores of L1-L4 at <-3.0 in DEXA bone density tests
* women with positive pregnancy tests before the trial or who planned to become pregnant within the following 3 years
* patients with a history of malignant tumor or malignant diseases (but the cases of cured disease with no relapse for the past 5 years were included in the present study)
* patients with abnormal blood potassium and phosphorus levels;
* patients with liver disease, kidney disease, respiratory disease, metabolic disease, or psychological disease;
* patients deemed to have less than 1-year life expectancy;
* patients with mental retardation or whose parents or legal guardians were older or had mental disabilities;
* other patients viewed as inappropriate by the staff

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Fusion rates | up to 5 year after operation
  This is assessed by postoperative computed tomography at 1 year after surgery

SECONDARY OUTCOMES:
Visual Analog Pain Scale (VAS) | 3, 6, and 12, months, and every year, up to 5 year after operation
  VAS is a measurement score that indicates pain severity status. VAS score comprised a 10-cm line with ''none'' (0) on one end of the scale and ''disabling pain'' (10) on the other.
Oswestry Disability Index (ODI) | 3, 6, and 12, months, and every year, up to 5 year after operation
  The ODI is based on a self-administered questionnaire measuring ''back-specific function.'' The questionnaire comprises 10 items, each with 6 levels of response. Each item is scored from 0 to 5, and the total summation is converted to a 0-100 scale.20 The ODI scores ranges from 0 to 100, with higher scores indicating severe symptoms.
EQ-5D | 3, 6, and 12, months, and every year, up to 5 year after operation
  EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
PainDETECT | 3, 6, and 12, months, and every year, up to 5 year after operation
  The painDETECT Questionnaire (PDQ) is a screening tool designed to detect neuropathic pain in patients with chronic low back pain (LBP) based on self-reported pain characteristics. The degree of the seven types of pain quality, the type of pain pattern, and the presence of radiating pain. From the three components of the PDQ, a total score is calculated; a high score indicates that the pain is likely to have a neuropathic component. Scoring is performed using a scoring manual, and results in a final screening score: a score of 0-12 indicates nociceptive pain, 19-38 indicates neuropathic pain, and 13-18 indicates mixed pain.
Fusion rates | every year, up to 5 year after operation
  This is assessed by postoperative simple radiography at 1 year after surgery
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | every year, up to 5 year after operation
  Device related adverse events (fracture, translation, subsidence, osteolysis), Surgery related adverse events (incidental durotomy, wound infection, re-operation, re-admission)

OTHER OUTCOMES:
Operation duration | Immediate after operation
  Intraoperative time
Intraoperative blood loss | Immediate after operation
  Intraoperative blood loss
Postoperative drainage | Within 3 days after operation
  Total drainage after surgery
Amount of transfusion | Within 7 days after operation
  Total transfusion during and after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyounggido, South Korea